CLINICAL TRIAL: NCT03756571
Title: Biomechanics and Walking in Cerebral Palsy: Ankle Foot Orthoses - Footwear Combinations
Brief Title: Cerebral Palsy: Ankle Foot Orthoses - Footwear Combinations
Acronym: CP-AFOFC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Orthocare Innovations (Industry); Hanger Clinic: Prosthetics & Orthotics (Other); Cascade Dafo (Industry)
Responsible Party: Principal Investigator, Kristie Bjornson, Associate Professor, Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21HD094823 (NIH)
Record Dates: First submitted 2018-11-05; First posted 2018-11-28 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Cerebral Palsy (CP)
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Study Design and Randomization. A randomized waitlist trial will be used to compare the AFO-FC to TSAFO in ambulatory children with CP.
Who Masked: Outcomes Assessor
Masking Description: Primary outcomes are Gait Profile Score (GPS), Gait Deviation Index (GDI), gait speed from three dimensional gait analysis and community walking activity are all collected via technology (three dimensional gait lab, accelerometry, thus masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ankle Foot Orthoses-Footwear Combination (Experimental): The intervention is a Ankle Foot Orthoses Footwear Combination (AFO-FC). This is some form of solid ankle AFO combined with modified footwear individually designed per algorithm.
  Interventions: Other: Ankle Foot Orthoses-Footwear Combination
- Traditional Solid Ankle AFO (TSAFO) (Active Comparator): The intervention is a solid AFO (SAFO) aligned with the ankle at 90 degrees and worn with regular footwear. We'll refer to this as the "traditional" SAFO (TSAFO)...
  Interventions: Other: Traditional Solid Ankle AFO (TSAFO)

INTERVENTIONS:
Other: Ankle Foot Orthoses-Footwear Combination — This is a solid AFO with angle of ankle in AFO and shoe modifications per algorithm based on physical exam and visual observation of lower extremity kinematics through stance phase of walking.
  Arms: Ankle Foot Orthoses-Footwear Combination
Other: Traditional Solid Ankle AFO (TSAFO) — This is a solid ankle AFO with angle of ankle in AFO at 90 degrees or neutral dorsiflexion/plantarflexion.
  Arms: Traditional Solid Ankle AFO (TSAFO)

SUMMARY:
Ambulatory children with cerebral palsy (CP) demonstrate altered lower limb biomechanical alignment in walking (e.g. excessive hip/knee flexion or equinus during stance) and experience walking activity limitations that negatively influence their ability to participate in day to day life. Ankle Foot Orthoses (AFO) are a fundamental rehabilitation strategy to facilitate walking in children with CP; yet, a review suggests that efficacy of the "traditional" solid AFO (TSAFO) in this population remains equivocal. A novel decision tree to guide orthotic prescription proposes a patient-specific method for adjusting AFO alignment and integrating footwear modifications (Ankle Foot Orthoses-Footwear Combinations, AFO-FC). This approach is based on visualizing the sagittal plane orientation of the ground reaction force vector with respect to lower limb segments during gait. The AFO-FC represents a paradigm shift in orthotic management as it accommodates ankle equinus contractures in a rigid AFO, reorients the tibial segment with a heel wedge under the AFO, and applies different heel, midsole and forefoot shoe modifications to restore lost ankle-foot rockers. The primary goal of AFO-FCs are to improve stability by facilitating more normal segment kinematics in single limb stance, decreasing hip/knee flexion. Despite their promise, evidence of an immediate positive effect on midstance alignment is limited, with no evidence of clinical effectiveness.

This proposal assesses the feasibility of using a randomized waitlist study to acquire pilot data on a targeted clinical cohort of children with CP evaluating the effectiveness of AFO-FCs as compared to TSAFO during daily life. Individual joint and combined kinematics and kinetics will be examined for potential mechanisms of action as well as daily walking performance, balance and satisfaction with the AFO-FC in 30 ambulatory children with CP, ages 4-9 years, with bilateral crouch or equinus gait pattern, comparing gait in TSAFO to the AFO-FCs.

DETAILED DESCRIPTION:
The goal of this proposal is to assess the feasibility of using a randomized waitlist study to acquire pilot data on a targeted clinical cohort of children with CP evaluating the effectiveness of AFO-FCs as compared to TSAFO during daily life. Individual joint and combined kinematics and kinetics will be examined for potential mechanisms of action as well as daily walking performance, balance and satisfaction with the AFO-FC in 30 ambulatory children with spastic diplegia CP, ages 4-9 years, with bilateral crouch or equinus gait pattern, comparing gait in TSAFO to the AFO-FCs.

Aim 1: Examine the effect of AFO-FC on individual joint kinematics, overall gait deviations and walking speed as compared to the TSAFO in children with CP. Multiple gait deviations (e.g. crouch or equinus) in CP result in slow, inefficient walking [14]. We hypothesize that the individualized ankle angle, leg segment alignment, and footwear profiles of the AFO-FCs will optimize lower limb joint kinematics, decrease overall gait deviations facilitating longer step lengths (improved stance stability), with resultant increased gait speed as compared to TSAFO. Instrumented gait analysis will assess gait speed and calculate changes in joint specific kinematics with the Gait Profile Score (GPS) and overall combined gait kinematics with the GDI.

Aim 2: Examine the effect of AFO-FC on daily walking activity, balance, mobility, and satisfaction as compared to the TSAFO in children with CP. We hypothesize that the AFO-FC will positively affect community walking activity levels, balance, physical activity and satisfaction as compared to the TSAFO. Walking activity will be captured by the StepWatch ® accelerometer; balance by the Pediatric Balance Scale; physical activity by the Patient Reported Outcomes Measurement System (PROMIS®) Pediatric Physical Activity and the Gait Outcomes Assessment List (GOAL); and satisfaction with device by the Orthotic and Prosthetic Users' Survey (OPUS).

ELIGIBILITY:
Inclusion Criteria:

* ambulatory children with spastic diplegia CP,
* spasticity primary movement disorder
* aged 4-9 years
* Gross Motor Function Classification System (GMFCS) levels of II or III
* clinically appropriate for a solid AFO based on physical exam/visual gait analysis criteria of:

  1. insufficient gastrocnemius length to allow knee extension with ankle dorsiflexion of 10 degrees and an uncompromised foot arch;
  2. low tone in the calf muscles with inability to control dorsiflexion during stance;
  3. insufficient calf muscle strength to prevent excessive dorsiflexion in stance and create a 'quasi stiff" ankle in terminal stance that allows the heel to rise from the ground; and
  4. insufficient triplanar boney stability of the foot during stance phase dorsiflexion

     Exclusion Criteria:
* Participants who have undergone:

orthopedic or neurological surgery less than 6 months prior to enrollment or injection therapies (phenol, botulinum toxin) less than 3 months prior to enrollment will be excluded.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristie F Bjornson, PhD, PT, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were approached and recruited through clinical care at Seattle Children's Hospital (SCH) or regionally by study team, once clinically deemed to meet inclusion criteria.
Pre-assignment Details: This was a randomized cross over design where those who randomized to TSAFO group first then crossed over without a washout period to the AFOFC treatment arm after 3 months of wearing the TSAFO.
Period: Overall Study
Arm/Group | Ankle Foot Orthoses-Footwear Combination | Traditional Solid Ankle AFO (TSAFO)
Started | 10 | 11
Completed | 9 | 10
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: These are the individual children who randomized to the two comparison conditions.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ankle Foot Orthoses-Footwear Combination | Traditional Solid Ankle AFO (TSAFO) | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Full Range); unit: years] | 7.3 [5.1 to 9.6] | 6.6 [4.2 to 9.8] | 6.9 [4.2 to 9.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 5 | 11
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline Gait Profile Score (GPS) at 3 Months-individual Lower Extremity Joint Kinematics
Description: The Gait Profile Score (GPS) represents the pattern of deviation as a single number and is derived from the same individual joint/limb gait kinematics as Gait Deviation Index (GDI) The GPS minimum value is 0 and maximum value is 20. A higher score is a worse outcome. An minimally clinically important difference is published to be 1.6 for children with CP.
Time Frame: 3 months post wearing assigned orthotic intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankle Foot Orthoses-Footwear Combination | Traditional Solid Ankle AFO (TSAFO)
Number analyzed (Participants) | 7 | 6
units on a scale | 0.41 (1.95) | -0.48 (1.47)
Statistical Analysis 1: Comparison: Ankle Foot Orthoses-Footwear Combination vs Traditional Solid Ankle AFO (TSAFO); Test type: Superiority; p = 0.36, t-test, 2 sided

2. Primary Outcome: Change in Right Baseline Gait Deviation Index (GDI) at 3 Months
Description: Gait Deviation Index (GDI) as a value representing overall gait deviation from a normal kinematic profile (0 to 120 scale) captures cumulative changes occurring at multiple joints and segments by side left/right. GDI has been shown to have concurrent validity with gross motor function and functional walking levels in children with CP. A score > 100 is considered in the normal range. A higher score is a better outcome.
Time Frame: 3 months post wearing assigned orthotic intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankle Foot Orthoses-Footwear Combination | Traditional Solid Ankle AFO (TSAFO)
Number analyzed (Participants) | 7 | 6
units on a scale | .07 (10.2) | 3.2 (5.8)
Statistical Analysis 1: Comparison: Ankle Foot Orthoses-Footwear Combination vs Traditional Solid Ankle AFO (TSAFO); Test type: Superiority; p = 0.50, t-test, 2 sided

3. Primary Outcome: Change in Baseline Walking Speed in Meters/Second (m/s) at 3 Months.
Description: Gait speed will be captured during the three dimensional gait analysis testing. Gait speed is measured in meters per second (m/sec) with range from 0 to ~ 3.0 m/sec for walking in children. A higher number of m/sec is considered a better outcome with minimally clinically important difference (MCID) of .10 m/s for persons with CP.
Time Frame: 3 months post wearing assigned orthotic intervention
Measure: Mean (Standard Deviation); unit: meters/second (m/s)
Arm/Group | Ankle Foot Orthoses-Footwear Combination | Traditional Solid Ankle AFO (TSAFO)
Number analyzed (Participants) | 7 | 6
meters/second (m/s) | -.03 (18) | .13 (.16)
Statistical Analysis 1: Comparison: Ankle Foot Orthoses-Footwear Combination vs Traditional Solid Ankle AFO (TSAFO); Test type: Superiority; p = 0.15, t-test, 2 sided

4. Primary Outcome: Change in Baseline Community Walking Activity Level at 3 Months in Strides/Day.
Description: Community walking activity will be captured by the ankle worn StepWatch ® accelerometer capturing change in average strides/day. The StepWatch ® is a two dimension accelerometer validated to capture when the foot leaves the ground for a metric of stride counts within the context of daily life. Average strides/day can range from 0 to unlimited strides/day. A higher number of strides/day is considered a better outcome.
Time Frame: 3 months post wearing assigned orthotic intervention
Measure: Mean (Standard Deviation); unit: strides/day
Arm/Group | Ankle Foot Orthoses-Footwear Combination | Traditional Solid Ankle AFO (TSAFO)
Number analyzed (Participants) | 9 | 10
strides/day | -804 (1131) | -182 (813)
Statistical Analysis 1: Comparison: Ankle Foot Orthoses-Footwear Combination vs Traditional Solid Ankle AFO (TSAFO); Test type: Superiority; p = 0.23, t-test, 2 sided

5. Primary Outcome: Change in Baseline Community Walking Intensity at 3 Months in Percent Time in High Stride Rates of > 60 Strides/Minute.
Description: Community walking activity will be captured by the ankle worn StepWatch Accelerometer capturing % time at high stride rates. Percent time at high stride rates (> 60 strides/min) can range from 0 to 100% with a higher percent considered a better outcome.
Time Frame: 3 months post wearing assigned orthotic intervention
Measure: Mean (Standard Deviation); unit: percentage of time in > 60 strides/min
Arm/Group | Ankle Foot Orthoses-Footwear Combination | Traditional Solid Ankle AFO (TSAFO)
Number analyzed (Participants) | 9 | 10
percentage of time in > 60 strides/min | -.03 (0.24) | -.15 (0.86)
Statistical Analysis 1: Comparison: Ankle Foot Orthoses-Footwear Combination vs Traditional Solid Ankle AFO (TSAFO); Test type: Superiority; p = 0.70, t-test, 2 sided

6. Primary Outcome: Change in Left Baseline Gait Deviation Index (GDI) at 3 Months
Description: Gait Deviation Index (GDI) as a value representing overall gait deviation from a normal kinematic profile (0 to 120 scale) captures cumulative changes occurring at multiple joints and segments by side LEFT/RIGHT. GDI has been shown to have concurrent validity with gross motor function and functional walking levels in children with CP. A score > 100 is considered in the 'normal' range. A higher score is a better outcome.
Time Frame: Change in Right baseline Gait Deviation Index (GDI) at 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankle Foot Orthoses-Footwear Combination | Traditional Solid Ankle AFO (TSAFO)
Number analyzed (Participants) | 7 | 6
units on a scale | -1.5 (2.7) | 1.3 (6.1)
Statistical Analysis 1: Comparison: Ankle Foot Orthoses-Footwear Combination vs Traditional Solid Ankle AFO (TSAFO); Test type: Superiority; p = 0.33, t-test, 2 sided

7. Secondary Outcome: Change in Balance From Baseline to 3 Months as Measured by Pediatric Balance Scale.
Description: The Pediatric Balance Scale (PBS) is a functional measure intended to assess balance in a clinical setting for children with neurological impairment. The PBS is a scaled scoring with range of 0 to 100 with a higher score a better outcome.
Time Frame: 3 months post wearing assigned orthotic intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ankle Foot Orthoses-Footwear Combination | Traditional Solid Ankle AFO (TSAFO)
Number analyzed (Participants) | 9 | 10
score on a scale | 12.8 (10.5) | 3.5 (5.8)
Statistical Analysis 1: Comparison: Ankle Foot Orthoses-Footwear Combination vs Traditional Solid Ankle AFO (TSAFO); Test type: Superiority; p = 0.03, Regression, Linear

8. Secondary Outcome: Change in Mobility From Baseline to 3 Months Change in Gait Outcome Assessment List (GOAL) Total Standard Score .
Description: Gait Outcomes Assessment List (GOAL) - The Gait Outcomes Assessment List (GOAL) is a outcome assessment to evaluate gait priorities and functional mobility for ambulant children with CP. The GOAL range of standard scores is 0 to 100 with a high score a better outcome. The GOAL will allow clinicians to better understand the motor abilities, priorities, and expectations of ambulant children with CP and to improve decision-making about appropriate interventions. The GOAL consists of 48 items grouped into seven domains: 1) activities of daily living and independence; 2) gait function and mobility; 3) pain, discomfort and fatigue; 4) physical activities, sports and recreation; 5) gait pattern and appearance; 6) use of braces and mobility aids; and 7) body image and self-esteem.
Time Frame: 3 months post wearing assigned orthotic intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ankle Foot Orthoses-Footwear Combination | Traditional Solid Ankle AFO (TSAFO)
Number analyzed (Participants) | 9 | 10
score on a scale | 7.91 (9.2) | -0.44 (5.5)
Statistical Analysis 1: Comparison: Ankle Foot Orthoses-Footwear Combination vs Traditional Solid Ankle AFO (TSAFO); Test type: Superiority; p = 0.03, Regression, Linear

9. Secondary Outcome: Difference Between Groups in Physical Function T-scores of Patient-Reported Outcomes Measurement Information System (PROMIS) After 3 Months Wearing Devices/Shoes.
Description: Parental report of Physical Function Mobility subscale T-scores from the Patient-Reported Outcomes Measurement Information System (PROMIS) pediatric survey. The PROMIS Physical Function subscale T score range is 0 to 100 with a higher score a better outcome. The mean of the T-score for Physical Function Mobility is 50 with a SD of 10, For parental report a score > or equal to 45 is consider Good, 36 - 44 Fair and < or equal to 35 Poor physical Function
Time Frame: 3 months post wearing assigned orthotic intervention
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Ankle Foot Orthoses-Footwear Combination | Traditional Solid Ankle AFO (TSAFO)
Number analyzed (Participants) | 9 | 10
T score | 36.2 (3.8) | 32.9 (3.9)
Statistical Analysis 1: Comparison: Ankle Foot Orthoses-Footwear Combination vs Traditional Solid Ankle AFO (TSAFO); Test type: Superiority; p = 0.08, t-test, 2 sided

10. Secondary Outcome: Difference Between Groups in Pain/Fatigue Level of the Gait Outcomes Assessment List (GOAL) After Wearing Devices/Shoes for 3 Months
Description: Parental report of pain/fatigue domain standard scores on the Gait Outcomes Assessment List (GOAL). The range of the pain/fatigue subscale of the GOAL 0 to 100. A higher score is a better outcome.
Time Frame: 3 months post wearing assigned orthotic intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ankle Foot Orthoses-Footwear Combination | Traditional Solid Ankle AFO (TSAFO)
Number analyzed (Participants) | 9 | 10
score on a scale | 88.3 (12.2) | 78.2 (16.7)
Statistical Analysis 1: Comparison: Ankle Foot Orthoses-Footwear Combination vs Traditional Solid Ankle AFO (TSAFO); Test type: Superiority; p = 0.18, t-test, 2 sided

11. Secondary Outcome: Difference Between Groups in Pain Interference After Wearing Devices/Shoes for 3 Months Pain Interference T Scores From PROMIS Pediatric Survey
Description: Parental report of selected pain and pain interference items from the Patient-Reported Outcomes Measurement Information System (PROMIS)pediatric survey. The Pediatric PROMIS pain interference subscale T score range is 0 to 100 with a lower score a better outcome. The mean is 50 with SD of 10. For the Pain interference a T score < 50 is considered within normal limits.
Time Frame: 3 months post wearing assigned orthotic intervention
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Ankle Foot Orthoses-Footwear Combination | Traditional Solid Ankle AFO (TSAFO)
Number analyzed (Participants) | 9 | 10
T score | 45.6 (8.6) | 53.4 (13.1)
Statistical Analysis 1: Comparison: Ankle Foot Orthoses-Footwear Combination vs Traditional Solid Ankle AFO (TSAFO); Test type: Superiority; p = 0.15, t-test, 2 sided

12. Secondary Outcome: Difference Between Groups in Satisfaction With Orthoses/Shoes After Wearing for 3 Months Per Orthotic and Prosthetic Users Survey (OPUS).
Description: Parental report of satisfaction raw score items from the Orthotic and Prosthetic Users' Survey (OPUS). The range of OPUS scores is 11-55 with a higher score a better outcome. The raw scores are employed as the survey validation for Rasch scores is not completed for children.
Time Frame: 3 months post wearing assigned orthotic intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ankle Foot Orthoses-Footwear Combination | Traditional Solid Ankle AFO (TSAFO)
Number analyzed (Participants) | 9 | 10
score on a scale | 42.1 (6.9) | 42.8 (4.7)
Statistical Analysis 1: Comparison: Ankle Foot Orthoses-Footwear Combination vs Traditional Solid Ankle AFO (TSAFO); Test type: Superiority; p = 0.80, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline consent visit through 3 month follow-up of initial randomized phase of trial and through the second cross over phase to the AFOFC condition.
Arm/Group | Ankle Foot Orthoses-Footwear Combination | Traditional Solid Ankle AFO (TSAFO)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 5/9 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ankle Foot Orthoses-Footwear Combination (N=9) | Traditional Solid Ankle AFO (TSAFO) (N=10)
Mild (Congenital, familial and genetic disorders) | 4 (7) | 5 (5) — inconvenience to day to day life (i.e. skin redness with device wear that lasts > 30 min post removal)
Moderate (Congenital, familial and genetic disorders) | 2 (3) | 6 (10) — required medical attention (i.e. Orthotist modified the device to address a blister resulting from wear of device)

LIMITATIONS AND CAVEATS:
Due to hardware failure in Dec 2020, there was a data loss of the gait outcomes at the OrthoCare Biomechanics Lab (gait lab). Thus the gait lab variables of GPS and GDI have a sample size of 13, where all other outcomes have a sample size of 19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT03756571/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT03756571/SAP_001.pdf